CLINICAL TRIAL: NCT00251407
Title: Phase I Study of Taxotere, Cisplatin, and CPT-11 in Advanced Solid Tumor Malignancies
Brief Title: Taxotere, Cisplatin, and CPT-11 in Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles S. Fuchs, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-149
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Solid Tumor
Keywords: Advanced solid tumor malignancy; cisplatin; CPT-11; taxotere
MeSH Terms: interventions — Docetaxel; Cisplatin; Irinotecan

ARMS (1):
- taxotere, cisplatin, irinotecan (Experimental)
  Interventions: Drug: Taxotere; Drug: Cisplatin; Drug: CPT-11

INTERVENTIONS:
Drug: Taxotere — Given intravenously on days 1 and 8 of a 21-day cycle. Participants can continue to receive study drug as long as there disease does not worsen and they do not experience serious side effects.
Drug: Cisplatin — Given intravenously on days 1 and 8 of a 21-day cycle. Participants can continue to receive study drug as long as there disease does not worsen and they do not experience serious side effects.
Drug: CPT-11 — Given intravenously on days 1 and 8 of a 21-day cycle. Participants can continue to receive study drug as long as there disease does not worsen and they do not experience serious side effects.

SUMMARY:
The purpose of this study is to find the highest dose of the combination of taxotere, cisplatin and CPT-11, that can be given without causing severe side effects. We also want to test the safety of this drug combination and see what effects (good and bad) it has on patients with advanced cancer for which there is no known curable treatment.

DETAILED DESCRIPTION:
* This is a Phase I clinical trial. We are unsure of the safest and most effective dose of the drugs and therefore are planning on treating 3-6 patients with a given dose before increasing to higher dose levels.
* Each patient will receive approximately two cycles of therapy. On day one and day eight, they will receive taxotere, cisplatin and CPT-11 intravenously. The cycle will begin again on day 22.
* The following tests and procedures will be performed: CAT scan prior to beginning therapy, after every 2 cycles of therapy, and at the end of the study; physical exam before each course of therapy; vital signs before and with each dose of therapy; routine blood tests before starting therapy and weekly during treatment; chest x-ray and echocardiogram before starting therapy and; toxicity assessment each week of therapy.
* Patients will remain on the study as long as their cancer responds to treatment and they do not have unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, incurable solid tumor malignancy
* 18 years of age or older
* ECOG performance status of < or = to 2
* Life expectancy of greater than 12 weeks
* WBC > 3,000/mm3
* ANC > 1,500/mm3
* Platelet count > 100,000/mm3
* Total bilirubin within normal limits
* SGOT < 2.5 x ULN
* Alkaline phosphatase < 4 x ULN

Exclusion Criteria:

* Prior chemotherapy for the treatment of metastatic or recurrent cancer
* Prior radiotherapy to greater than or equal to 15% of bone marrow
* Prior pelvic radiation therapy
* Prior nitrosoureas or mitomycin C
* Myocardial infarction in the past 6 months
* Major surgery in past 2 weeks
* Uncontrolled serious medical or psychiatric illness
* Uncontrolled diarrhea
* Peripheral neuropathy > grade 1
* Pregnant or lactating women
* Clinically apparent central nervous system metastases or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1999-09; Primary Completion 2003-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose of weekly taxotere, cisplatin and CPT-11 in patients with incurable solid tumor malignancies. | 3 years

SECONDARY OUTCOMES:
To define the dose-limiting toxicities of the combination of drugs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Fuchs, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Enzinger PC, Ryan DP, Clark JW, Muzikansky A, Earle CC, Kulke MH, Meyerhardt JA, Blaszkowsky LS, Zhu AX, Fidias P, Vincitore MM, Mayer RJ, Fuchs CS. Weekly docetaxel, cisplatin, and irinotecan (TPC): results of a multicenter phase II trial in patients with metastatic esophagogastric cancer. Ann Oncol. 2009 Mar;20(3):475-80. doi: 10.1093/annonc/mdn658. Epub 2009 Jan 12. PMID 19139178